CLINICAL TRIAL: NCT05448222
Title: Effect of Sarcopenia on the Efficacy and Prognosis of HCC Treated With Systemic Therapies
Brief Title: Effect of Sarcopenia on Hepatocellular Carcinoma(HCC) After Systemic Therapies
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Eastern Hepatobiliary Surgery Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Gang Chen, MD, Clinical Professor, Principal Investigator, First Affiliated Hospital of Wenzhou Medical University
Other Study IDs: sarcopenia and liver cancer
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Hepatocellular Carcinoma; Sarcopenia
Keywords: hepatocellular carcinoma; sarcopenia; prognosis; adverse events; systemic therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Sarcopenia | interventions — Tomography, X-Ray Computed; Hand Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: gait speed; ct scan; grip strength and chair stand test — The chair stand test was administered, and the time required for the patient to stand five times from a sitting position without using the arms was measured. CT scan was to scan the patient's third lumbar level. For the gait speed test, the time that patients spent walking 8 meters on a flat indoor floor at usual walking speed was measured.Grip strength test:the dominant hand and the nondominant hand were measured twice intermittently (kg), and the average value of 4 values was obtained.

SUMMARY:
Sarcopenia is associated with the prognosis of HCC and cholangiocarcinoma. But there has been rare study focusing on the effect of sarcopenia on the prognosis of HCC treated with systemic therapy, such as interventional therapy, targeted therapy, chemotherapy and immunotherapy and so on.

DETAILED DESCRIPTION:
By tracking the short-term and long-term results of HCC patients treated with systemic therapy,the difference of short-term results between patients with sarcopenia and patients without sarcopenia was analyzed, and the correlation between sarcopenia and short-term and long-term results of patients after systemic treatments was explored, so as to improve people's awareness of sarcopenia and pay attention to its prevention and treatment.All implementation details are based on the newest EuropeanWorking Group on Sarcopenia in Older People(EWGSOP) definition. The investigators consecutively admitted patients the questionnaire and evaluated the assessment of muscle strength (grip strength test and chair stand test), muscle quantity (L3 plane total skeletal muscle area) and physical performance (gait test) following the F-A-C-S approach, to confirm patients with sarcopenia accurately. And by tracking the short-term and long-term outcomes, the differences were analyzed and the relationship between sarcopenia and prognosis of systemic treatments was explored.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of hepatocellular carcinoma
* No cancer other than liver cancer has been diagnosed
* Age ≥18 years
* child-pugh score≤7

Exclusion Criteria:

* uncompleted standard tests and questionnaires
* received other therapies
* Patients who had other causes of muscle weakness (injury, fracture, stroke, etc.)
* Patients who missing CT data or CT scan did not reach the level of the third lumbar vertebra (L3)
* lost follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical diagnosis of hepatocellular carcinoma admitted to the first affiliated hospital of wenzhou medical university and received standard tests and questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
complications | 3 months
  The complications were classified according to the Clavien-Dindo classification, such as hypertension, fever, abdominal pain and so on.
overall survival | 2 years
  Overall survival was defined as the time from initiation of lenvatinib to death for any reason.
progression free survival | 2 years
  Progression free survival was defined as the time from initiation of lenvatinib to first progression or death.

SECONDARY OUTCOMES:
Hospital stay | 3 months
  The time that patients spent in the hospital was recorded.
Hospital cost | 3 months
  Hospital cost that patients spent was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Gang Chen, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith C, Woessner MN, Sim M, Levinger I. Sarcopenia definition: Does it really matter? Implications for resistance training. Ageing Res Rev. 2022 Jun;78:101617. doi: 10.1016/j.arr.2022.101617. Epub 2022 Apr 1. PMID 35378297
- [Background] Leong DP, Teo KK, Rangarajan S, Lopez-Jaramillo P, Avezum A Jr, Orlandini A, Seron P, Ahmed SH, Rosengren A, Kelishadi R, Rahman O, Swaminathan S, Iqbal R, Gupta R, Lear SA, Oguz A, Yusoff K, Zatonska K, Chifamba J, Igumbor E, Mohan V, Anjana RM, Gu H, Li W, Yusuf S; Prospective Urban Rural Epidemiology (PURE) Study investigators. Prognostic value of grip strength: findings from the Prospective Urban Rural Epidemiology (PURE) study. Lancet. 2015 Jul 18;386(9990):266-73. doi: 10.1016/S0140-6736(14)62000-6. Epub 2015 May 13. PMID 25982160
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Kobayashi A, Kaido T, Hamaguchi Y, Okumura S, Shirai H, Yao S, Kamo N, Yagi S, Taura K, Okajima H, Uemoto S. Impact of Sarcopenic Obesity on Outcomes in Patients Undergoing Hepatectomy for Hepatocellular Carcinoma. Ann Surg. 2019 May;269(5):924-931. doi: 10.1097/SLA.0000000000002555. PMID 29064889
- [Background] Dasarathy S, Merli M. Sarcopenia from mechanism to diagnosis and treatment in liver disease. J Hepatol. 2016 Dec;65(6):1232-1244. doi: 10.1016/j.jhep.2016.07.040. Epub 2016 Aug 8. PMID 27515775